CLINICAL TRIAL: NCT03494829
Title: Physical Activity, Motor Competence, Pulmonary Function, and Quality of Life in Children With Severe Spinal Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Johan Kibsgård, Senior Consultant, Oslo University Hospital
Other Study IDs: OUHRH
Record Dates: First submitted 2017-03-15; First posted 2018-04-11 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Scoliosis; Idiopathic, Infantile; Scoliosis; Juvenile; Scoliosis Neuromuscular; Scoliosis in Neurofibromatosis; Scoliosis; Congenital, Postural; Scoliosis in Skeletal Dysplasia; Scoliosis Associated With Other Conditions; Scoliosis; Congenital, Due to Bony Malformation; Scoliosis
Keywords: early onset scoliosis; motor competence; physical activity; pulmonary function; health related quality of life
MeSH Terms: conditions — Scoliosis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Observation study about physical activity, motor competence, pulmonary function, and health related quality of life in children, surgically treated for early onset scoliosis

DETAILED DESCRIPTION:
Early Onset Scoliosis (EOS) defines patients who develop deformities of the spine and/or thorax in the embryologic development or in the early childhood. The exact prevalence of EOS in Norway is unknown, but it is assumed to be approximately 200-300 new EOS patients every year. EOS is a severe condition, whereby some of the most common and also most severe consequences of the deformity are severe pulmonary problems. The patients may require extensive orthopedic treatment from early childhood and until maturity to avoid serious consequences with severe pulmonary problems and shortening of life.

EOS' secondary problems, including severe consequences on the pulmonary function might contribute to enhanced inactivity. Inactivity contributes to further negative impact on development of the musculoskeletal system, motor competence and pulmonary function. Considering the severity of EOS and children's reduced life expectancy, it is extremely important that EOS children achieve the favorable impact of physical activity during their growth. Insufficient level of activity might worsen the prognosis, thus counteracting the treatment's ambitions. The investigator's aim is to extend the knowledge about level of activity, motor competence, pulmonary function, and health related quality of life in Norwegian children, surgically treated for EOS.

ELIGIBILITY:
Inclusion Criteria:

* Early onset scoliosis diagnosis
* Understand and speak Norwegian
* For physical activity test: Walking ability
* For motor competence test and/or pulmonary function test: Ability to understand the test and cooperate

Exclusion Criteria:

* Other spinal disease, not early onset scoliosis

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children treated at the Norwegian National Unit for Surgical Treatment of Non-malignant Pathologies in Pediatric Spine, Oslo University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Physical Activity, assessed by use of accelerometer | Change in activity counts from baseline to activity counts at 6 months and 12 months.
  Physical Activity will be measured objective by use of an accelerometer (used over 7 days), recorded as Activity Counts/ minutes

SECONDARY OUTCOMES:
Airway resistance, assessed by use of plethysmography | Change in measures from baseline and to 12 months
  Children >8 years will also be assessed by use of plethysmography. Airway resistance will be measured, recorded as the ratio of driving pressure divided by flow through the airways
Pulmonary residual volume and total lung capacity, assessed by use of plethysmography | Change in measures from baseline and to 12 months
  Children >8 years will also be assessed by use of plethysmography. Residual volume (liters) and total lung capacity (liters) will be measured.
Pulmonary function, assessed by use of diffusion capacity test | Change in measures from baseline and to 12 months
  Children >8 years will be assessed by use of diffusion capacity test. Diffusing capacity or transfer factor of the lung for carbon monoxide (CO) (DLCO) will be measured.
Pulmonary function, assessed by use of spirometry | Change in measures from baseline and to 12 months
  All participants will go through spirometry. Vital capacity (VC), Forced vital capacity (FVC), Forced expiratory volume (FEV) at timed intervals of 0.5, 1.0 (FEV1), 2.0, and 3.0 seconds and maximal voluntary ventilation (MVV) will be measured (liters)
Forced expiratory flow, assessed by use of spirometry | Change in measures from baseline and to 12 months
  All participants will go through spirometry. Forced expiratory flow 25-75% (FEF 25-75) will be measured (liters/second)
Motor competence, assessed by use of Movement Assessment Battery of Children- 2. edition | Baseline and after 12 months
  Motor competence will be assessed by use of Movement Assessment Battery of Children- 2. edition
Health related quality of life in children | Change in parents answers of health related quality of life of their child from baseline, to 6 months and to 12 months.
  Health related quality of life will be assessed by use of the Early Onset Scoliosis 24-item Questionnaire (EOSQ-24). Total score, ranged 0 (worst) to 100 (best), including 11 subdomain scores, ranged 0 (worst) to 100 (best) will be calculated.
Health related quality of life in adolescents | Change in subjective answers of health related quality of life from baseline, to 6 mounts and to 12 mounts.
  Among participants > 16 years, health related quality of life will be assessed by use of the Scoliosis Research Society 22- item (SRS-22) questionnaire. Total score and 5 subdomain scores, all ranged 5 (best) to 1 (worst), will be calculated.
Shoulder function | Baseline and after 12 months
  A physiotherapist will assess the active shoulder range of motion, categorized as normal, active range of motion >50% of perceived motion, or active range of motion <50% of perceived motion. shoulder flexion, extension, abduction, and rotation will be measured.
Physical Activity, assessed by use of questionnaire | Change in subjective answers of everyday activity from baseline, to 6 mounts and to 12 mounts.
  Physical Activity will be subjective measured by use of a questionnaire regarding participants' everyday activity. Participants range their activity in several sports activities from never (1) to several days a week (4).The questionnaire is previous used in a national survey study regarding physical activity among children and adolescents in Norway.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Johan Kibsgård, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No